CLINICAL TRIAL: NCT00817401
Title: Effect of Systemic Hypothermia on Neonatal Hypoxic-Ischemic Encephalopathy
Brief Title: Systemic Hypothermia Improves Outcome of Hypoxic-Ischemic Encephalopathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhengzhou University (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Professor Changlian Zhu, Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HN-200084001
Record Dates: First submitted 2009-01-02; First posted 2009-01-06 (Estimated); Last update posted 2009-01-06 (Estimated); Status verified 2009-01

CONDITIONS: Hypoxic-Ischemic Encephalopathy
Keywords: asphyxia; hypothermia; hypoxic-ischemic encephalopathy; neonates
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Asphyxia; Hypothermia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: hypothermia — For the systemic hypothermia treatment (TS Med 200, Germany), the infants were nursed under an open unit, covered only by a diaper and a thin linen, loosing heat to the environment and to a cooling mat¬tress which was perfused by circulating liquid at a variable temperature. The rectal temperature was targeted at 33.5 °C (range of 33 to 34 °C) and was meant to be achieved within 60 min. The body temperature was checked every 10 min during induction hypothermia and every hour during the remaining period of cooling. The duration of hypothermia was 72 hrs. Rewarming was started by stopping the cooling system. The infant was meant to reach a 36.5°C rectal temperature in 6 hrs after stopping cooling to prevent rebound hyperthermia.
  Other Names: TS Med 200, Germany

SUMMARY:
Perinatal asphyxia-induced brain injury is one of the most common causes of morbidity and mortality in term and preterm neonates. Birth asphyxia accounts for 23% of neonatal deaths globally and survivors suffer from long term neurological disability and impairment. Although many neuroprotective strategies appeared promising in animal models, most of them were not feasible and effective in human newborns. However, hypothermia was reported not to be effective if introduced beyond and thus should be introduced within 6 hrs after birth.Applying this selection criterion naturally would deprive many patients of the opportunity of hypothermia treatment.

DETAILED DESCRIPTION:
Hypoxic-ischemic encephalopathy of the newborn infant remains a significant socio-economic health problem worldwide. Moderate to severe HIE of newborn infants is associated with a high rate of death or long-term disabilities. Historically, treatment has been purely supportive including stabilizing cardio-respiratory functions and treating convulsions. Recent multi-center trials assessing the effects of hypothermia demonstrated improved outcome in term neonates with moderate hypoxic-ischemic encephalopathy (HIE). However, hypothermia was not effective beyond 6 hrs after brain injury. The aim of this study was to investigate whether systemic hypothermia induced up to 10 hrs after birth would improve the neurodevelopmental outcome at 18 months in infants with moderate or severe HIE.

ELIGIBILITY:
Inclusion Criteria:

1. Gestation age ≥37 weeks and body weight >2500g.
2. with one of the following factors:

   1. Apgar score<5 at 5min;
   2. Assisted respiration >3min due to respiratory distress;
   3. pH≤7.1 of cord or arterial blood within 60min after birth;
   4. clinical manifestation of encephalopathy during the first 10 hrs of life.

Exclusion Criteria:

1. Major congenital abnormalities;
2. Head trauma or skull fracture causing major intracranial hemorrhage;
3. Mild HIE;
4. Financial problems of the parents;
5. Lack of permanent address;
6. Postnatal age > 10 hrs

Ages: 1 Hour to 10 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2002-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Mortality and disability rate. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Changlian Zhu, MD, PhD, Study Director — Zhengzhou University
Locations (1):
- NICU, the Third Affiliated Hospital, Zhengzhou University, Zhengzhou, Henan, China